CLINICAL TRIAL: NCT03447197
Title: Five-year Patency of No-touch Saphenous Vein Grafts in On-pump Versus Clamp-less Off-pump Coronary Artery Bypass Surgery: A Sub-study of a Multicenter Randomized Controlled Trial
Brief Title: Five-year Patency of No-touch Saphenous Vein Grafts in On-pump Versus Clamp-less Off-pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Ninos Samano M.D., Consultant in Cardiothoracic Surgery, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLL-689991
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Stenoses
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-Pump (Active Comparator): Use of extracorporeal circulation
  Interventions: Procedure: The use of extracorporeal circulation
- Off-Pump (No Intervention)

INTERVENTIONS:
Procedure: The use of extracorporeal circulation — The use or not of extracorporeal circulation during the coronary artery bypass procedure.
  Arms: On-Pump

SUMMARY:
Randomised controlled trials (RCTs) have shown high long-term patency for no-touch saphenous vein grafts (NTSVGs), comparable to the internal thoracic artery in on-pump coronary artery bypass grafting (CABG). RCTs on patency in NTSVGs in off-pump CABG have not been published yet. Orebro University Hospital participated in the CABG Off- or On-pump Revascularization study (CORONARY, ClinicalTrials.gov number, NCT00463294) and included fifty-six patients. Accordingly, this is a sub-study and the aim was to assess the midterm patency in NTSVGs in clamp-less off-pump versus on-pump CABG at five-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they:

  1. provided written informed consent;
  2. were >21 years of age;
  3. required isolated CABG with median sternotomy;
  4. had at least one of the following risk factors:

     1. had peripheral vascular disease (previous peripheral bypass, amputation or anklebranchial index <0.90),
     2. had cerebrovascular disease (history of stroke, transient ischemic attach or carotid stenosis ≥70%),
     3. had renal insufficiency (creatinine above upper limit of normal),
     4. were ≥70 years of age, or
     5. were between the ages of 60-69 with one of the following: i. had diabetes and taking an oral hypoglycemic agent and/or insulin, ii. required urgent revascularization (i.e., waiting in hospital for revascularization after an acute coronary syndrome), iii. were a recent smoker (within 1 year of randomization), or iv. had left ventricular ejection fraction ≤35%, OR
     6. were between the ages of 55-59 with two of the following: i. Diabetes and taking an oral hypoglycemic agent and/or insulin, ii. required urgent revascularization (i.e., waiting in hospital for revascularization after an acute coronary syndrome, iii. were a recent smoker (within 1 year of randomization), or iv. had a left ventricular ejection fraction ≤35%

Exclusion Criteria:

* Patients were excluded if they:

  1. required a concomitant cardiac procedure associated with CABG;
  2. had a contraindication to off-pump or on-pump CABG (e.g., calcified aorta, intramuscular left anterior descending artery, calcified coronaries, small target vessels);
  3. had a concomitant life-threatening disease likely to limit life expectancy to less than 2 years;
  4. were previously enrollment in the CORONARY Trial;
  5. required emergency CABG surgery (i.e., immediate revascularization for hemodynamic instability); OR
  6. required a redo CABG.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Graft patency | Five years postoperatively
  Graft patency as assessed with computed tomography angiography